CLINICAL TRIAL: NCT05771077
Title: The Effect of Poly Amido Amine Dendrimer, Nano-hydroxyapatite and Their Combination on Micro Hardness of Demineralized Enamel and Their Clinical Efficacy in Management of White Spot Lesions
Brief Title: Effect of Poly Amido Amine Dendrimer, Nano-hydroxyapatite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asmaa Khater
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — Poly(amidoamine); Dendrimers; nano-hydroxyapatite-collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients have White spot lesions (Experimental): White spot lesions (WSLs) are defined as enamel surface and subsurface demineralization, without cavitation. These manifestations represent the first clinical observation of the progression of dental caries, with the possibility of being reversed
  Interventions: Drug: Poly(Amidoamine) dendrimer

INTERVENTIONS:
Drug: Poly(Amidoamine) dendrimer — to evaluate the Remineralizing effect of Poly Amido Amine Dendrimer, Nanohydroxy apatite & Their Combination on demineralized enamel & Their Clinical Efficacy on White Spot lesion
  Other Names: Nano-hydroxyapatite

SUMMARY:
Dental caries is a common oral disease. The process of caries formation is a cycle of remineralization and demineralization with various stages being either reversible or irreversible.

DETAILED DESCRIPTION:
White spot lesions (WSLs) are defined as enamel surface and subsurface demineralization, without cavitation. These manifestations represent the first clinical observation of the progression of dental caries, with the possibility of being reversed.

WSLs are characterized by a white, chalky, opaque appearance and are commonly located in pits, fissures, and smooth surfaces of teeth. However, after the placement of fixed orthodontic appliances, there are an increasing number of plaque retention sites due to the presence of brackets, bands, wires and other applications, which make oral hygiene more difficult, and limit naturally occurring self-cleansing mechanisms. As a consequence, there is an increased risk of demineralization and, conclusively, of WSLs forming on smooth surfaces, if there is no effective plaque removal

The clinical characteristics of these lesions include loss of normal translucency of the enamel because of altered light properties with a chalky white appearance, particularly when dehydrated; a fragile surface layer susceptible to damage from probing, particularly in pits and fissures; increased porosity, particularly of the subsurface, with increased potential for uptake of stains; reduced density of the subsurface, which may be detectable radiographically, with transillumination or with modern laser detecting devices; and potential for remineralization, with an increased resistance to further acid challenge particularly with the use of enhanced remineralization treatments.

It is possible to find numerous therapies for WSLs, for instance, hygiene education, fluorides, phosphopeptide compounds, xylitol and infiltrative resins, microabrasion and/or bleaching, and preparation and restoration. The professional application or prescription of fluorides for home use includes: gels, toothpastes, mouthwashes and varnishes. The fluoride ions are revealed in three ways: sodium monofluorophosphate, sodium fluoride and amine fluoride. It has been found that high fluoride concentrations promote WSL remineralization However; it occurs in the enamel surface and inhibits the ions' movement through the subsurface, affecting the subsurface remineralization and therefore, the light reflection

ELIGIBILITY:
Inclusion Criteria:

* The patients have at least 3 WSLS.
* The patients aged between 16 and 25 years old
* The patients with good general health and no systemic disease.

Exclusion Criteria:

* Presence of enamel hypoplasia or dental fluorosis.
* Presence of carious cavity.
* Allergy to fluoride gel being used in this stufy
* Patients who have a significant medical history, including pregnancy and breast feeding and smokers.
* Patients who have evidence of reduced salivary flow or significant tooth wear.
* Patients who had participating in concurrent clinical trials or who had recently participated in other clinical trials of an investigational drug or device.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Remineralization | 3 months
  to evaluate the Remineralizing effect of Poly Amido Amine Dendrimer and Nanohydroxy apatite alone or combined on demineralized enamel on White Spot lesion. Remineralization will be assessed by radiodensity using digital radiography

CONTACTS AND LOCATIONS:
Overall Officials: Wael Essam Gamel, Professor, Study Chair — Al-Azhar Faculty of Dentistary for girls
Locations (1):
- Faculty of Dentistary - Al-Azhar University, Cairo, Egypt